CLINICAL TRIAL: NCT02900820
Title: Safety of Discontinuing Patient Antibiotic Treatment When Physicians no Longer Consider it Necessary
Brief Title: Safety of Discontinuing Patient Antibiotic Treatment
Acronym: STOP-AB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Society of Family and Community Medicine (Other)
Responsible Party: Principal Investigator, Carl Llor, Principal Investigator, Spanish Society of Family and Community Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/101
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2020-10

CONDITIONS: Infectious Diseases; Respiratory Tract Infections
Keywords: Anti-Bacterial Agents; Primary Health Care; Drug Resistance, Microbial; Respiratory Tract Infections
MeSH Terms: conditions — Communicable Diseases; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Novel intervention group (Experimental): Discontinuing antibiotic therapy.
  Interventions: Other: Discontinuing antibiotic therapy
- Usual intervention group (Experimental): Usual strategy of continuing antibiotic treatment.
  Interventions: Other: Continuing antibiotic therapy

INTERVENTIONS:
Other: Discontinuing antibiotic therapy — Patients assigned to this group will be asked to discontinue antibiotic therapy.
  Arms: Novel intervention group
Other: Continuing antibiotic therapy — Patients assigned to this group will be asked to complete antibiotic therapy.
  Arms: Usual intervention group

SUMMARY:
There is no evidence that discontinuing antibiotic therapy for non-bacterial infections is safe. The main objective of this study is to determine whether discontinuation of antibiotic therapy when a clinician no longer considers it necessary makes any difference in terms of the number of days with severe symptoms. This is a multicentre, open-label, randomised controlled clinical trial. The study will be conducted in ten primary care centres in Spain. We will include patients from 18 to 75 years of age with uncomplicated acute respiratory tract infections (RTIs) in whom: antibiotics are not necessary; or those diagnosed with clinical conditions for which antibiotics might be necessary but according to the history and clinical examination the physician considers that antibiotics are not needed or the patient feels that the antibiotic regimen has not worked as expected; or several doses of an antibiotic have been taken from leftovers found in the household or obtained at the pharmacy without any medical prescription for a clinical condition for which antibiotics are not necessary. The patients will be randomly assigned to the usual strategy of continuing antibiotic treatment (usual intervention group) or discontinuing antibiotic therapy (novel intervention group). A sample size of 215 patients per group was calculated on the basis of a reduction of one day in the duration of severe symptoms as a clinically relevant outcome. The primary outcome will be duration of severe symptoms, i.e. symptoms scored 5 or 6 by means of a symptom diary. Secondary outcomes will include: antibiotics taken, adverse events, patient satisfaction, and complications within the first 3 months.

DETAILED DESCRIPTION:
Introduction: General practitioners (GP) have always been told to continue an antibiotic regimen once the patient has initiated it in order to prevent the patient from acquiring resistant microorganisms. This might be true for confirmed bacterial infections; however, continuing an antibiotic regimen when this is not indicated might hasten the acquisition of resistant organisms and cause adverse events. Since 2011 the Spanish Society of Family Medicine has been recommending GPs to ask their patients to stop taking antibiotics when they suspect a viral infection. However, there is no evidence that discontinuing antibiotic therapy for these conditions is safe. The main objective of this study is to determine whether discontinuation of antibiotic therapy when a GP no longer considers it necessary makes any difference in terms of the number of days with severe symptoms.

Methods: This is a multicentre, open-label, randomised controlled clinical trial. The study will be conducted in ten primary care centres in Spain. We will include patients from 18 to 75 years of age with uncomplicated acute respiratory tract infections (RTIs) in whom: 1. Antibiotics are not necessary; or 2. Those diagnosed with clinical conditions for which antibiotics might be necessary but according to the history and clinical examination the GP considers that antibiotics are not needed or the patient feels that the antibiotic regimen has not worked as expected; or 3. Several doses of an antibiotic have been taken from leftovers found in the household or obtained at the pharmacy without any medical prescription for a clinical condition for which antibiotics are not necessary. The patients will be randomly assigned to the usual strategy of continuing antibiotic treatment (usual intervention group) or discontinuing antibiotic therapy (novel intervention group). A sample size of 215 patients per group was calculated on the basis of a reduction of one day in the duration of severe symptoms as a clinically relevant outcome. The primary outcome will be duration of severe symptoms, i.e. symptoms scored 5 or 6 by means of a symptom diary. Secondary outcomes will include: antibiotics taken, adverse events, patient satisfaction, and complications within the first 3 months. A post-trial implementation observational clinical study by means of a qualitative analysis is planned to be carried out after the clinical trial to know the percentage of the use of the strategy of discontinuing antibiotic treatment and the pros and cons of its use.

Ethics and dissemination: The study was approved by the Ethical Board of Fundació Jordi Gol i Gurina (reference number: 16/093) and informed consent will be obtained from all the patients included. The findings of this trial will be disseminated through research conferences and peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria: Patients with uncomplicated respiratory tract infections [common cold, influenza, pharyngitis, rhinosinusitis, acute bronchitis, and acute exacerbations of mild-to-moderate chronic obstructive pulmonary disease] who has previously taken any dose of antibiotic due to any of the following 3 clinical scenarios and accepts to participate in the clinical trial will be included:

* Patients diagnosed with clinical conditions for which antibiotics are not necessary;
* Patients diagnosed with a clinical condition for which antibiotics might be necessary but according to the history and clinical examination the primary health physician considers that antibiotics are not needed to be taken or the patients feel that the antibiotic regimen has not worked as expected and feel they need clinical reassessment
* Patients who have taken some doses of an antibiotic (from leftovers found in the household or obtained at the pharmacy without any medical prescription) for a clinical condition for which antibiotics are not necessary

Exclusion Criteria:

* Subjects under 18 and over 75 years of age
* Patients with confirmed bacterial infection
* Patients requiring hospital admission
* Severe impairment of signs (impairment of consciousness, respiratory rate > 30 respirations per minute, heart rate > 125 beats per minute, systolic blood pressure < 90 mm Hg, diastolic blood pressure < 60 mm Hg, temperature > 40°C, oxygen saturation < 92%)
* Problems to comply with treatment at home - sociopathy or psychiatric problems, drug or alcohol addiction, or within an inadequate family setting -
* Lack of tolerance to oral treatment, such as the presence of nausea and vomiting, gastrectomy, post-surgery and/or diarrhoea
* Significant comorbidity, including severe renal failure, hepatic cirrhosis, severe heart failure, immunosuppression - chronic HIV infection, transplantation, neutropenic, or patients receiving immunosuppressive drugs or corticosteroids -
* Terminal disease
* Admitted to a long-term residence
* Difficulty to attend the programmed visits
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-01; Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Duration of severe symptoms | From 14 to 28 days after the index visit
  Days with symptoms scoring 5 or 6 by means of a six-point Likert scale

SECONDARY OUTCOMES:
Adverse effects of the medication | From index visit to 28 days after the initial visit
  Any adverse effect appearing from day 0 to 28
Antibiotic consumption | From index visit to day 28
  Any antibiotic taken by the patient
Satisfaction with health care by means of a questionnaire | Day 28 after the index visit
  Satisfaction degree stated by the patient at day 28
Belief in the effectiveness of antibiotic therapy by means of a questionnaire | Day 28 after the index visit
  Degree of patient's belief in how effective antibiotics are for uncomplicated respiratory tract infections
Rate of complications | Within the first 3 months
  Any complication related to the uncomplicated respiratory tract infection within the 3 first months after the index visit

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Cots, Professor, Study Director — University of Barcelona
Locations (5):
- Spain (5):
  - Coll d'en Rabassa Primary Health Center, Palma de Mallorca, Balearic Islands
  - Manso - Via Roma Primary Care Center, Barcelona, Catalonia
  - La Marina Primary Care Center, Barcelona, Catalonia
  - Guinardó Primary Care Center, Barcelona, Catalonia
  - Jaume I Primary Care Center, Tarragona, Catalonia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gilbert GL. Knowing when to stop antibiotic therapy. Med J Aust. 2015 Feb 16;202(3):121-2. doi: 10.5694/mja14.01201. No abstract available. PMID 25669463
- [Background] Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. BMJ. 2010 May 18;340:c2096. doi: 10.1136/bmj.c2096. PMID 20483949
- [Background] Dekker AR, Verheij TJ, van der Velden AW. Inappropriate antibiotic prescription for respiratory tract indications: most prominent in adult patients. Fam Pract. 2015 Aug;32(4):401-7. doi: 10.1093/fampra/cmv019. Epub 2015 Apr 24. PMID 25911505
- [Background] Morgan DJ, Okeke IN, Laxminarayan R, Perencevich EN, Weisenberg S. Non-prescription antimicrobial use worldwide: a systematic review. Lancet Infect Dis. 2011 Sep;11(9):692-701. doi: 10.1016/S1473-3099(11)70054-8. Epub 2011 Jun 12. PMID 21659004
- [Background] Goossens H, Ferech M, Vander Stichele R, Elseviers M; ESAC Project Group. Outpatient antibiotic use in Europe and association with resistance: a cross-national database study. Lancet. 2005 Feb 12-18;365(9459):579-87. doi: 10.1016/S0140-6736(05)17907-0. PMID 15708101
- [Derived] Llor C, Moragas A, Bayona C, Cots JM, Hernandez S, Calvino O, Rodriguez M, Miravitlles M. Efficacy and safety of discontinuing antibiotic treatment for uncomplicated respiratory tract infections when deemed unnecessary. A multicentre, randomized clinical trial in primary care. Clin Microbiol Infect. 2022 Feb;28(2):241-247. doi: 10.1016/j.cmi.2021.07.035. Epub 2021 Aug 4. PMID 34363942
- [Derived] Llor C, Moragas A, Bayona C, Cots JM, Molero JM, Ribas J, Fothy JF, Gutierrez I, Sanchez C, Ortega J, Arranz J, Botanes J, Robles P. The STOP-AB trial protocol: efficacy and safety of discontinuing patient antibiotic treatment when physicians no longer consider it necessary. BMJ Open. 2017 Jun 6;7(5):e015814. doi: 10.1136/bmjopen-2016-015814. PMID 28592581